CLINICAL TRIAL: NCT00477932
Title: Human Disease With Mutation of Nonmuscle Myosin Heavy Chain Genes
Brief Title: Genes Mutation Pentalogy of Cantrell
Status: Withdrawn | Type: Observational
Why Stopped: Physician's chose to not follow through with the study.
Sponsor: Children's Healthcare of Atlanta (Other)
Collaborators: Emory University (Other); University of Texas Southwestern Medical Center (Other); University of California, San Francisco (Other); Ben-Gurion University of the Negev (Other); Brigham and Women's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital and Health System Foundation, Wisconsin (Other); University of Puerto Rico (Other)
Responsible Party: Sponsor
Other Study IDs: 182-2006
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Pentalogy of Cantrell; Mutations in Non-muscle Genes
Keywords: Pentalogy of Cantrell; mutations; DNA; RNA
MeSH Terms: conditions — Pentalogy of Cantrell

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will collect blood, urine, and other tissue samples from 50 patients study-wide with Pentalogy of Cantrell and other inherited diseases that involve mutations in non-muscle genes. Mutations in non-muscle genes have been shown to result in human defects involving blood platelets, kidney, hearing and sight. The major objective of this protocol is to study a variety of blood, tissue and urine samples by looking at protein, DNA, and RNA in those collected samples.

DETAILED DESCRIPTION:
Pentalogy of Cantrell is a very rare disorder in which patients have a combination of severe defects of the middle of the chest including the sternum (breastbone), diaphragm (muscle which separates the chest from the abdomen), heart, and abdominal wall. The defects can affect both males and females and is apparent at birth or shortly after.

This study will collect blood, urine, and other tissue samples from 50 patients study-wide with Pentalogy of Cantrell and other inherited diseases that involve mutations in non-muscle genes. Mutations in non-muscle genes have been shown to result in human defects involving blood platelets, kidney, hearing and sight. The major objective of this protocol is to study a variety of blood, tissue and urine samples by looking at protein, DNA, and RNA in those collected samples.

Enrollment in this study is entirely voluntary and the subject can elect to withdraw from the study at any time. Each subject will receive an oral and written explanation of this study and the purpose, procedures, and risks of this study in language that is comprehensible. The Investigator will be available to answer any questions the subject may have regarding the study. If the subject is a minor, the parent who signs the consent for the minor must be the legally recognized parent or guardian. Where deemed appropriate, the child will also be included in all discussions about the trial and a minor's assent will be obtained. The parent or guardian will sign on the designated line on the informed consent attesting to the fact that the child had given assent. If the minor child refuses to provide assent, then participation in the study will not occur. Informed consent will be obtained by the Investigator or designee, and a copy of the signed consent document will be given to the subject and placed in the subject's medical record. Subjects may withdraw permission of use of blood/tissue/urine specimens at any time.

Tissue and/or blood and/or urine samples from participating institutions that have identified cases of Pentalogy of Cantrell and/or related syndromes will be collected. These samples will be sent to the National Heart, Lung, and Blood Institute (NHLBI) for analysis and kept for a period of 5 years, unless the subject withdraws permission during that period. Standard methods will be used to collect the blood, tissue, and/or urine samples. For example, blood samples will be obtained from routine blood drawing and tissue may be obtained from previously obtained tissue secondary to surgery.

Samples that are sent to the NHLBI for analysis will have identifiers on them, so if new information is discovered, the research subject may be contacted. All samples will be stored in a locked storage facility to maximize patient confidentiality.

Anticipated Adverse Events are listed in the protocol and consent. Unanticipated Adverse Events will be reported to the appropriate institutions. All serious adverse events will be reported by the Investigator verbally and in writing to the Clinical Director and the NHLBI IRB within the time frame set by the protocol. The nature of this study does not warrant a DSMB, therefore the principal Investigator, Dr. Robert Adelstein will provide oversight of the safety and data analysis of the conduct of this study.

The benefit of this study is discovery of the disease and the mutation that causes the disease, therefore yielding generalizable knowledge regarding the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Those patients who have Pentalogy of Cantrell (as defined under STUDY DESIGN) or other diseases that could involve mutation of any of the nonmuscle myosin genes that will be defined in future amendments
* Outside Institutions- All ages will be included
* At the Clinical Center-Those subjects that are > 2 years of age and older

Exclusion Criteria:

* screening for subjects who may be asymptomatic, but who could be carrying the gene
* we will exclude all children under the age of 2

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Those patients who have Pentalogy of Cantrell (as defined under STUDY DESIGN) or other diseases that could involve mutation of any of the nonmuscle myosin genes that will be defined in future amendments
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
•Those patients who have Pentalogy of Cantrell (as defined under STUDY DESIGN) or other diseases that could involve mutation of any of the nonmuscle myosin genes that will be defined in future amendments | Undetermined

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Heiss, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] A literature search regarding this disease or condition was performed by the NHLBI Informationalist, Mary Ryan, NIH Library. The 5 key words utilized for this literature search were: nonmuscle myosin II, myosin II mutation, midline defects, Pentalogy of Cantrell, and Thoracoabdominal Syndrome. Please see attached sheets